CLINICAL TRIAL: NCT06665074
Title: Inflammatory Challenge in Human Aggression.
Acronym: LPSS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emil Coccaro, Professor of Psychiatry, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023H0217; R01MH133925-01A1 (NIH)
Record Dates: First submitted 2024-10-21; First posted 2024-10-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Intermittent Explosive Disorder
Keywords: IED; Inflammation; Cytokines; Aggression
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Inflammation; Aggression | interventions — Endotoxins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo (saline infusion)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aggressive Subjects (Experimental): Subjects with Intermittent Explosive Disorder (IED)
  Interventions: Biological: Endotoxin (E. coli O:113, Reference Endotoxin); Other: Saline (Placebo)
- Non-Aggressive Subjects (Other): Subjects without IED
  Interventions: Biological: Endotoxin (E. coli O:113, Reference Endotoxin); Other: Saline (Placebo)

INTERVENTIONS:
Biological: Endotoxin (E. coli O:113, Reference Endotoxin) — Dosage of endotoxin is 0.8 ng/Kg body Weight
Other: Saline (Placebo) — Volume of saline to be the same as volume of endotoxin

SUMMARY:
The goal of this clinical trial is to explore the differences in behavioral and cytokine response to a low dose infusion of endotoxin (vs. placebo) in individuals with histories of frequent, problematic, impulsive aggression ("aggressives") compared to similar individuals without this history ("controls"). Endotoxin is a substance that produces a reliable inflammation response in human subjects. The main questions it aims to answer are:

* Do aggressive individuals have greater self-rated anger responses to low-dose endotoxin compared with controls?
* Do aggressive individuals have greater analog aggressive responses (in the Taylor Aggression Paradigm) to low-dose endotoxin compared with controls?
* Do aggressive individuals have greater hostile attributional and negative emotional responses (in the V-SEIP) to low-dose endotoxin compared with controls?
* Do aggressive individuals have greater plasma pro-inflammatory responses to low-dose endotoxin compared with controls?
* Do aggressive individuals display a greater activation of brain responses to anger-related picture during an MRI scan during low-dose endotoxin compared with controls? Researchers will compare endotoxin to a placebo (a look-alike substance that contains no drug) explore the differences in behavioral and cytokine response to a low dose infusion of endotoxin (vs. placebo) in individuals with histories of frequent, problematic, impulsive aggression ("aggressives") compared to similar individuals without this history ("controls").

Participants will:

* Receive a low-dose of endotoxin and placebo on two (2) separate days. The study drugs will be given through a plastic tube inserted in a forearm vein.
* Visit the laboratory on at least two (2) separate days to receive the endotoxin and placebo.
* Complete rating forms, behavioral testing, and an MRI on each of the two (2) laboratory days.

DETAILED DESCRIPTION:
While elevations of circulating pro-inflammatory modulators correlate directly with variables of aggression, and direct application of cytokines to specific cortico- limbic regions in animals elicit aggressive responding, no studies have tested the hypothesis that acute increases in pro-inflammatory modulators can/will increase aggressive behavior in humans. The investigators aim to demonstrate a causal relationship between pro-inflammatory cytokines and aggression in human subjects by showing that an acute pro-inflammatory state, via endotoxin challenge, will increase aggressive responding, anger ratings, and hostile social cognition, to a greater degree in "aggressive" (n = 45), compared with "non-aggressive" (n = 45), individuals with mood/anxiety/ stress-related and/or personality disorders. The proposed study is a double-blind comparison of endotoxin/placebo challenge in the same individuals (within-subject) as a function of aggression status. Aggressive individuals will have high lifetime aggression (> 12 on Life History of Aggression: LHA) and be positive for an average of two anger attacks per week and/or three anger attacks per year that include physical assault of another person and/or or non-trivial destruction of property. "Non-Aggressive" individuals will be similar diagnostically but will have low lifetime aggression. "Aggressive responding" will be assessed using the Taylor Aggression Paradigm (TAP), "Anger" will be assessed by self-reported assessments (Profile of Mood States: POMS), and "Hostile Social Cognition" will be assessed by the Video-Social and Emotional Information Processing (V-SEIP) paradigm. The primary plasma pro-inflammatory outcome measures will be a composite of CRP, IL-6, IL-8, and TNF-α (as in the investigators' previous studies). MRI scans will including task-based scans involving "explicit" and "ambiguous" social threat. The investigators hypothesize that aggressive responding, anger ratings, and hostile social cognition (Primary Outcomes) and Composite Plasma Pro-Inflammatory Marker levels (Secondary Outcome), will be greater after endotoxin, compared with placebo, and will be greater in "aggressive" than "non- aggressive" study participants. The Investigators also hypothesize that these variables will correlate with dimensional measures of aggression. In addition, the investigators hypothesize that amygdala responses to explicit social threat (anger faces) will be enhanced (greater BOLD fMRI signal response) after Endotoxin, and that cortico-limbic responses to ambiguous social threat (V-SEIP) will be reduced (i.e., lesser BOLD fMRI signal response) in all study participants but reduced to a greater extent in "aggressive", compared with "non- aggressive", study participants. Finally, the investigators hypothesize that the pro-inflammatory effects of the endotoxin challenge will result in reduced connectivity between the functional edges supporting higher aggressive behavior and that endotoxin challenge will facilitate stronger connections among nodes associated with low aggressive behavior. If supported, this study will provide a strong rationale for clinical trials of anti-inflammatory agents in impulsive aggressive individuals.

ELIGIBILITY:
Inclusion Criteria:

"Aggressive Subjects" will have a current DSM-5 diagnosis of Intermittent Explosive Disorder (IED) and have a Life History of Aggression (LHA) > 12.

"Control Subjects" will not have current or past history of IED and will have LHA scores < 11 ("Control Subjects" may have a past, but not current, history of Major Depression (MD), Generalized Anxiety Disorder (GAD), Panic Disorder (PDx), or Post-Traumatic Stress (PTSD) Disorder.

Participant is between 21 and 55 years of age and is able to give informed consent.

Participant is physically healthy as confirmed by medical history, physical evaluation, and (in females) a negative pregnancy test.

Exclusion Criteria:

Participants with a current clinically significant medical condition.

Participants current co-morbid Major Depression (MD), Generalized Anxiety Disorder (GAD), Panic Disorder (PDx), or Post-Traumatic Stress (PTSD) Disorder.

Participants currently taking prescribed medications for an active medical or psychiatric condition.

Participants not free of prescribed medications for four weeks.

Participants with Grade 2 or higher abnormalities on clinical laboratory examination (e.g., CBC with Differential, Metabolic Panel, and PT/INR/PTTa).

Participants with Bradycardia (i.e., heart rate < 50 beats/minute) or other Grade 2 or higher ECG abnormality.

Participants with autoimmune conditions (e.g., asthma, psoriasis, etc.)

Participants who are immunocompromised.

Participants taking immunomodulatory, or anti-inflammatory, agents.

Participants that are pregnant, breastfeeding, or plan to become pregnant within nine months of enrollment in the study.

Female study participants of childbearing potential must remain abstinent or agree to use a highly effective form of contraception (e.g., an intrauterine device). Childbearing potential is defined as, study participants who have reached menarche and have not undergone a documented sterilization procedure (i.e., hysterectomy, bilateral oophorectomy, or salpingotomy), and have not reached menopause.

Life history of bipolar disorder / schizophrenia / organic mental syndrome, or intellectual disability.

Current alcohol / drug use disorder of greater than mild severity.

Current suicidal ideation.

History of a suicide attempt in the past year prior to study entry.

Life history of > 3 or more suicide attempts of any type.

Life history of any moderately severe suicide attempt.

Current or life history of homicidal ideation.

Current or life history of felony assault and/or battery.

Currently on parole for aggressive behavior.

Allergy, or contraindication, to receiving endotoxin.

Current treatment with opiates or any agents that affect pain threshold (exclusionary for the TAP).

Unwilling/unable to sign informed consent document.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) - Anger | Before and during the Endotoxin/Placebo Infusion for up to six hours only on ach of the two study days..
  Self-report questionnaire of "anger". Scale goes form 0-48 with higher scores meaning greater anger.

SECONDARY OUTCOMES:
Taylor Aggression Paradigm (TAP) | Done once during the endotoxin (and placebo) infusion only. The TAP takes about 30 minutes.
  An analog assessment of aggression widely used in human studies of aggression. This is the number of times that a selection of higher and very-high shock was set by the subject against the "confederate".
Video-Social Emotional Information Processing (V-SEIP) | Done one during the endotoxin (and placebo) infusion only. The V-SEIP takes about 30 minutes on each of the two study days..
  A computer-delivered task that assesses hostile attributional bias and negative emotional response to ambiguous social threat. The scores range from 0-3 with the higher numbers mean the more hostile attribution and negative emotional response.
Pro-Inflammatory Cystokines (IL-6, THN-Alpha) | Prior to and after infusion of endotoxin and placebo for up to six hours only on each of the two study days.
  These are pro-inflammatory cytokines that are stimulated for release by endotoxin. These values range from 0 to > 100 with the higher values representing greater inflammation.
Functional MRI | Once during the Endotoxin Infusion and once during the Salin Infusion only. The MRI scan takes 90 minutes on each of the two study days.
  BOLD Signal Response to Explicit (Anger Faces), and to Ambiguous, Social Threat.

CONTACTS AND LOCATIONS:
Overall Officials: Emil F. Coccaro, MD, Principal Investigator — The Ohio State University College of Medicine
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identifed data will be shared.
Time Frame: Start date: Only after the study is completed and data analysis has been completed.
Access Criteria: University faculty at US and International Institutions. Only de-identified data will be released as data files.